CLINICAL TRIAL: NCT04399603
Title: Multi-organ Failure in SARS-CoV2: Identifying Mechanisms and Potential Therapeutic Targets
Brief Title: Mechanisms of Multi-organ Failure in COVID-19
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 283783
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID critically unwell patients
- Non-Covid critically unwell Patietns
  Interventions: Other: no intervention-mechanistic study

INTERVENTIONS:
Other: no intervention-mechanistic study — no intervention-mechanistic study
  Groups: Non-Covid critically unwell Patietns

SUMMARY:
In the United Kingdom, there are currently 138,000 confirmed patients with coronavirus, causing 18,738 deaths. Whilst the disease may be mild in the majority of patients, a significant proportion of patients require intensive care therapy and a ventilator due to lung injury. In addition to lung injury/failure (acute respiratory distress syndrome (ARDS)), around 50% of patients admitted to intensive care develop acute kidney injury (AKI) (requiring advanced support via haemofiltration) and multi-organ failure.

It is unclear why patients suffering from COVID-19 develop such severe lung injury (requiring life support or ventilation) or indeed why patients develop other organ dysfunction such as kidney injury. The investigators hypothesis that this may due to an over-reaction of the immune system particularly in the lungs. This then results in the release of various mediators and biological messengers which can be pushed into the blood bloodstream (exacerbated by positive pressure generated by the ventilator). These mediators then travel, via the blood, to other organs such as the kidney where they cause inflammation and injury of cells, resulting in organ failure.

The investigators would like to apply their well-established laboratory methods to further the scientific community's knowledge of this severe and deadly viral condition and we hope that this would lead to the development of medication that would treat this deadly virus.

DETAILED DESCRIPTION:
COVID-19 is a highly contagious virus, causing a global health emergency. A significant number (~17%) of hospitalised patients become severely unwell and require admission to an intensive care unit (ICU) due to lung failure (acute respiratory distress syndrome (ARDS)) and multi-organ failure (MOF). Sadly, 51.8% of COVID-ARDS patients develop kidney failure, which has a markedly increased risk of dying (61%). We have learned that kidney failure starts several days after lung failure, which suggest an initial viral "attack" on the lungs followed by kidney involvement several days later.

Cytokines are "signalling" molecules made by cells, which in healthy individuals help fight disease. It was initially thought that in COVID-19, lung cells release excessive cytokines (i.e. cytokine storm), which then cause kidney injury and MOF. However, research has demonstrated that cytokine levels in blood are actually very low and not enough to explain the extent of organ injury in COVID-19. This perhaps explains why treatment strategies aimed at specifically damping down the action of these particular cytokines in COVID-19 have failed. Consequently, there remains no cure for COVID-19 MOF, and whilst treatments such as steroids, manage symptoms, have a general anti-inflammatory effect and improve mortality, 30% of intensive care patients still die. Therefore, urgent research is needed to improve scientific knowledge of this condition and identify new therapies.

Microvesicles (MVs) are extremely small particles released by cells and carry various chemicals including cytokines, from inside the cell, packaged securely and safely within membranes (cellular envelopes). These vesicles act as 'postmen' delivering chemical messengers (e.g. cytokines) between cells and are important in various diseases where inflammation is implicated. The investigators have demonstrated that MVs have a fundamental role in the development of organ failure in laboratory models of non-COVID ARDS but the investigators do not yet know the role of these vesicles in the development of ARDS/MOF in COVID-19.

The investigators hypothesise that during COVID-19 infection of the lung, significant numbers of MVs are released within the lung (especially in severe COVID-19), which then "transmit" signals and inflammation to other organs via the bloodstream, causing organs to fail. Furthermore, as chemical messengers (e.g. cytokines) are hidden inside these vesicles, they are not measured by standard laboratory techniques and may explain why there are low cytokine levels in blood. This may also clarify why treatments inhibiting circulating cytokines (not hidden in vesicle membranes) have failed.

To explore these ideas, the group aim to investigate MVs in blood and urine of ICU patients with severe COVID-19 (20mls blood (1 1/3 tablespoons); 10ml urine (3/4 tablespoon)). The investigators intend to examine which chemicals are present in these tiny vesicles and to relate this information to the clinical progress or otherwise of patients. These data will help the scientific community understand the chemical systems involved in severe COVID-19, tell us the significance of MVs and whether blocking MV signalling could lead to new treatments for COVID-19. Furthermore, analysis of these MVs may allow the investigators to identify patients who are likely to become seriously ill, which would help in planning treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-90 years;
* Patients diagnosed with COVID-19 and without COVID-19 (control purposes);
* Patients who have developed evidence of organ injury failure (requiring oxygen).

Exclusion Criteria:

* Patients who are under the age of 18;
* Refusal to consent/gain assent;
* Presence of an advanced directive to withhold or to withdraw life-sustaining treatment;
* Moribund patient likely to die within 24 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically unwell patients requiring organ support
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation in inflammatory mediators in patients with multi-organ failure suffering from COVID-19 | 18 months
  This will involve measurement of microvesicles in blood (numbers of MVs per µL)
Variation in inflammatory mediators in patients with multi-organ failure suffering from COVID-19 | 18 months
  This will involve measurement of microvesicles in bronchoalveolar lavage fluid (numbers of MVs per µL)
Variation in inflammatory mediators in patients with multi-organ failure suffering from COVID-19 | 18 months
  This will involve measurement of microvesicles in urine (numbers of MVs per µL)

SECONDARY OUTCOMES:
Correlation of inflammatory mediators in the bronchoalveolar lavage fluid with extent of lung injury (e.g. based upon oxygen requirement) | 18 months
  The aforementioned inflammatory markers will be correlated with level fo lung injury which will be based upon the level of oxygen required by patients. (numbers of MVs per µL)
Correlation of circulating inflammatory mediators with renal and cardiovascular markers | 18 months
  The aforementioned inflammatory markers will be measured in renal outcomes (creatinine and urine output) and cardiovascular markers (e.g. natriuretic peptides (BNP and NT pro-BNP) and Troponin). (numbers of MVs per µL)
Assess the role of inflammatory mediators obtained from patients in the development of renal injury using in vitro | 18 months
  models (i.e. applying these inflammatory mediators isolated from these clinical samples on kidneys cells in a petri dish) (numbers of MVs per µL)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Imperial College NHS Trust, London

IPD SHARING:
Plan to Share IPD: No